CLINICAL TRIAL: NCT02331472
Title: The Efficacy of Urine Biomarker in Patient With Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: The Efficacy of Urine Biomarker in Patient With Interstitial Cystitis/Painful Bladder Syndrome (Pilot Study)
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Soo Choo, Professor, Asan Medical Center
Other Study IDs: 2014-1220
Record Dates: First submitted 2015-01-01; First posted 2015-01-06 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Chronic Interstitial Cystitis
Keywords: interstitial cystitis; biomarker
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — RNA in urine specimen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Interstitial cystitis: Patients who have been diagnosed with interstitial cystitis/bladder pain syndrome. The group includes both patients with or without Hunner lesion on cystoscopy
- Control: Adult participants without history of interstitial cystitis/bladder pain syndrome

SUMMARY:
This study is to evaluate the efficacy of urine biomarker in patients with interstitial cystitis/painful bladder syndrome

ELIGIBILITY:
Inclusion Criteria:

1. must have experienced bladder pain, urinary urgency and frequency for at least 6 months prior to entry into the study
2. Pain VAS >4
3. PUF score >13
4. ICQ score >12

4) cystoscopic record within 2years

Exclusion Criteria:

1. Patients who are pregnancy or, childbearing age without no contraception
2. Patient with microscopic hematuria, if not excluded that no evidence of neoplastic tumor examination
3. patients with urine culture showing evidence of urinary tract infection 1month prior to the study
4. Accompanied medical problem below

   * Tuberculosis in urinary system
   * Bladder cancer, urethral cancer, Prostate cancer
   * Recurrent cystitis
   * Anatomical disorder
5. Patients had prior surgery (bladder augmentation, cystectomy)
6. Patients with neurologic disorder
7. Patients with indwelling catheter or intermittent self-catheterization
8. Patients with psychological problem

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Interstitial cystitis
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2016-01-14 (Actual); Study Completion 2016-01-14 (Actual)

PRIMARY OUTCOMES:
Difference of RNA expression of the urine biomarker between the interstitial cystitis and control groups | 1day
  Difference of RNA expression of the urine biomarker between the interstitial cystitis and control groups

SECONDARY OUTCOMES:
Difference of RNA expression of the urine biomarker between Hunner ulcer interstitial cystitis and non-ulcer interstitial cystitis groups | 1day
  Difference of RNA expression of the urine biomarker between Hunner ulcer interstitial cystitis and non-ulcer interstitial cystitis groups
Difference of RNA expression of the urine biomarker in interstitial cystitis according to pain score on the visual analogue scale | 1day
  Difference of RNA expression of the urine biomarker in interstitial cystitis according to pain score on the visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Asan medical center Institutional review board, Seoul

IPD SHARING:
Plan to Share IPD: No